CLINICAL TRIAL: NCT06102486
Title: Speech Perception in Noise as an Improved Marker for Neurocognitive Dysfunction
Brief Title: MCI Speech in Noise
Status: Recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Christopher E. Niemczak, Research Scientist, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02002079
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCI: Participants diagnosed with or suspected to have MCI
- Control: Participants without MCI

SUMMARY:
The purpose of this study is to determine whether people with MCI (Mild Cognitive Impairment) and healthy comparison subjects differ with respect to their ability to hear soft sounds and how their brain understands and processes sound. The investigators are also evaluating, within those with MCI, whether the hearing tests are associated with neurocognitive functioning. The investigators are interested in learning whether changes in cognition in those with MCI can be detected using tests of how the brain processes sound. The investigators hypothesize that participants with MCI will score worse on both hearing tests and neurocognitive tests than participants without MCI. Participants are asked to complete multiple types of hearing tests, take a series of neurocognitive tests, and complete a few questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with or suspected to have MCI (for MCI group) or are cognitively normal (for Control group)
* Absence of other risk factors that might affect CAP (Central Auditory Processing) performance (e.g., active ear infections, congenital developmental delay, severe hearing loss)
* Age 55-80
* Normal hearing sensitivity (<40 dB HL Pure Tone Average (average of 500, 1000, 2000 Hz) thresholds bilaterally
* Normal middle ear function defined by tympanometry (0.3-2.0 ml)
* Native English speaker

Exclusion Criteria:

* Active ear infections or abnormal middle ear pathology
* Other health condition prohibiting the completion of the CAP test battery
* Mild to profound peripheral hearing loss (>40 dB (decibel) HL (hearing loss) Pure Tone Average (average of 500, 1000, 2000 Hz) bilaterally
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* History of CNS (Central Nervous System) disorder that might severely impact cognitive function (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis, neurosyphilis, intracranial tumors, history of significant head trauma with loss of consciousness (≥30 min), and cerebrovascular disease)
* Severe mental illness (e.g., schizophrenia, bipolar disorder)
* Current, uncontrolled medical condition that could affect cognition (e.g., hypertension)
* History of substance use disorder within the (other than nicotine/caffeine)
* Non-correctable severe hearing or vision loss
* Use of "Cognition Enhancing Drugs"
* Frequent, severe headaches (occasional headaches or migraines are fine)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The community in and around Lebanon, NH and patients from DHMC.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-18 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Hearing-in-Noise Test Performance | 1 time point (takes 15 minutes)
  The performance for Hearing in Noise Tests (HINT) between energetic masking and 2-talker informational masking (IM). Performance will be measured by the lowest signal-to-noise ratio (volume at which sentences are presented compared to background noise volume) that can be heard by the participant.
Triple Digit in Noise Test Performance | 1 time point (takes 15 minutes)
  Performance for the behavioral Triple Digit (TDT) between energetic masking and 2-talker informational masking (IM). Performance will be measured by the lowest signal-to-noise ratio (volume at which digits are presented compared to background noise volume) that can be heard by the participant.
Size of auditory neural response in background noise | 1 time point (takes 45 minutes)
  The change in amplitude of neural response between energetic masking and 2-talker informational masking (IM).
Timing of auditory neural response in background noise | 1 time point (takes 45 minutes)
  The change in latency of neural response between energetic masking and 2-talker informational masking (IM).

CONTACTS AND LOCATIONS:
Locations (1):
- Space Medicine Lab at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States